CLINICAL TRIAL: NCT01607424
Title: Specific Versus General Cognitive Remediation for Schizophrenia
Brief Title: Specific Cognitive Remediation for Schizophrenia
Acronym: RECOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Centre hospitalier Saint Jean de Dieu - ARHM (Other); Saint Anne's Hospital (Other)
Responsible Party: Principal Investigator, Nicolas FRANCK, Pr, Professor (Claude Bernard University), head of department (Hôpital le Vinatier), principal investigator, Hôpital le Vinatier
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECOS
Record Dates: First submitted 2012-05-11; First posted 2012-05-30 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia
Keywords: cognitive rehabilitation; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RECOS: 42 hours CR, 14 week-treatment. (Experimental): RECOS(Cognitive Remediation for Schizophrenia) exercises were designed by SBT Company and adapted by Vianin et al (2007) for specific use in schizophrenia. It includes computer based and paper and pencil exercises that target 5 main cognitive functions. RECOS modules focus on the relevant cognitive domains, which have been recommended by the MATRICS consensus. Each exercise has 10 difficulty levels. Allocation of the training modules in RECOS was determined according to the standard scores obtained in the comprehensive neuropsychological assessment. Each patient participated in the module corresponding to his/her most altered cognitive area.
  Interventions: Behavioral: cognitive remediation
- CRT: 42 hours CR, 14 week-treatment (Active Comparator): CRT (Cognitive Remediation Therapy) exercises are the ones used by Wykes et al (1999). The CRT method consists of 3 modules: flexibility, memory (A and B) and planning (A and B). Each module involves a series of paper and pencil exercises with parallel forms providing with gradual difficulty.
  Interventions: Behavioral: cognitive remediation

INTERVENTIONS:
Behavioral: cognitive remediation — RECOS: cognitive remediation for schizophrenia CRT: cognitive remediation therapy

SUMMARY:
Rationale:

Cognitive deficits are a core feature in schizophrenia. Conventional treatments (antipsychotic medication and psychological treatments) have limited effects so cognitive remediation programs were designed to alleviate the problems. Interventions typically involve a variety of exercises in a paper and pencil or a computerized format with a growing number of specialized computer programs now being developed. However, many of these programs lack specificity which does not allow an individual's specific needs to be addressed. More targeted interventions might increase the effects of therapy so RECOS - COgnitive REmediation for Schizophrenia - was developed to fit this gap.

Methods: This is a multicenter, randomized, controlled study comparing patients aged 18 to 45 years suffering from schizophrenia according to DSM-IV-TR. RECOS will be compared to an already validated program (CRT).

220 patients will be randomized as follows :

* Arm 1 : RECOS (42 h)
* Arm 2 : CRT (42 h) The recruitment is performed by psychiatrists in Lyon, Paris, Clermont-de-l'Oise, Niort, Bordeaux, Ville-Evrard and Lausanne.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 to 45 years
* French speaker or French schooling since 7 years
* clinical stability
* diagnosis of schizophrenia

Exclusion Criteria:

* visual or auditory disorder
* history of neurological illness or trauma
* alcohol or drug dependence
* mental retardation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in executive functioning at week 12 | week 12
  BADS(Behavioral Assessement of Dysexecutive Functions) total score

SECONDARY OUTCOMES:
Change from baseline in executive functioning, attention, memory and visuospatial abilities at week 12 | week 12
  comprehensive neuropsychological assessment
Change from baseline in symptoms at week 12 | week 12
  PANSS (Positive And Negative Symptoms Scale)
Change from baseline in self-esteem at week 12 | week 12
  Rosenberg scale
Change from baseline in insight at week 12 | week 12
  Birchwood scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Franck, Principal Investigator — Hôpital le Vinatier

REFERENCES:
- [Result] Franck N, Duboc C, Sundby C, Amado I, Wykes T, Demily C, Launay C, Le Roy V, Bloch P, Willard D, Todd A, Petitjean F, Foullu S, Briant P, Grillon ML, Deppen P, Verdoux H, Bralet MC, Januel D, Riche B, Roy P; Other members of the Cognitive Remediation Network; Vianin P. Specific vs general cognitive remediation for executive functioning in schizophrenia: a multicenter randomized trial. Schizophr Res. 2013 Jun;147(1):68-74. doi: 10.1016/j.schres.2013.03.009. Epub 2013 Apr 9. PMID 23583327